CLINICAL TRIAL: NCT04623697
Title: Covid-19 and Type 1 Diabetes - a Multicenter Study
Brief Title: Covid-19 Infection and New Onset Type 1 Diabetes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Collaborators: Steno Diabetes Center Odense (Other); Steno Diabetes Center Nordjylland (Other); Aarhus University Hospital (Other); Steno Diabetes Center Sjaelland (Other Government); Steno Diabetes Center Copenhagen (Other)
Responsible Party: Principal Investigator, Claus Bogh Juhl, MD., Ph.D., Clinical Professor, Esbjerg Hospital - University Hospital of Southern Denmark
Other Study IDs: S-20200119
Record Dates: First submitted 2020-11-09; First posted 2020-11-10 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Covid19; type1diabetes
Keywords: Covid19; Type 1 diabetes
MeSH Terms: conditions — COVID-19; Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Blood for research biobank
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Although recognized as an autoimmune disease the etiology of type 1 diabetes remains unknown. Virus infections has been suggested as a possible agent triggering the autoimmune reaction finally resulting in beta-cell destruction and fate of insulin secretion. SARS Cov-2 virus enters the infected cells by binding to the ACE-2 receptor, which is abundant in many tissues including the pancreas. Accordingly, SARS Covid-19 infection may trigger the development of type 1 diabetes either by an activation of the immune system or directly via beta-cell infection and destruction.

Our aim is to study the impact of the Covid-19 epidemic on the development of type 1 diabetes. This will be done in two ways: a clinical study and an epidemiological follow up. During the next two years, adult patients with newly diagnosed type 1 diabetes will be asked to participate. Type 1 diabetes will be diagnosed by usual means and a mixed meal tolerance test will be performed at time of diagnosis and after one year to evaluate beta-cell function. People with type 1 diabetes and serologically documented previous SARS Covid-19 will be compared with people with no previous infection regarding beta-cell function and fate of insulin secretion. In addition, we will estimate the number of new diagnosed type 1 diabetes patients compared to previous years.

DETAILED DESCRIPTION:
Background

Although recognized as an autoimmune disease, the etiology of type 1 diabetes mellitus (T1D) remains undetermined. One dominant hypothesis is that a recent virus infection elicits or enhances an autoimmune reaction, resulting in CD4+ and CD8+ T-cells recognizing pancreatic antigens and subsequently targeting the beta-cells of the pancreas. This results in a gradual but irreversible loss of beta-cell function.

Various enterovirus species have been suspected as causative factors of T1D. However, many different viruses may carry the potential to induce T1D via one of the above-mentioned mechanisms, including respiratory infections.

Most people are presently immunologically inert to SARS-Cov-2, but a large proportion of the world's population is expected to be infected over the next few years, with the global focus having now shifted to slowing the spread (1). The pandemic of COVID-19 therefore provides an opportunity to study a possible correlation between a novel type of virus infection and the development of T1D.

Aim

Our overall aim is to study the impact of Covid-19 on the incidence and the phenotype (beta-cell function at time of diagnosis and at follow up) of newly diagnosed adult patients with T1D in a multicenter study, with enrolments to occur in both Denmark and Portugal.

Method

The following study populations are established over a two-year period, beginning in October 2020:

1. Study population 1: Newly diagnosed adult patients with T1D according to usual practice, stratified for the presence of SARS-Cov-2-antibodies (+/-), in both Denmark and Portugal.
2. Study population 2: A control population of the same age (+/- 3 years) and sex from each participant country, potentially from the national blood banks. This will provide the SARS-Cov-2 status of the background population. Each newly diagnosed T1D patient is matched with five control persons.

Study 1: Clinical study: Study 1:

Inclusion criteria:

* T1D patients diagnosed according to standard practice (including Hba1c, C-peptide, presence of GAD (or islet-cell) antibodies).
* Patient is attending a hospital unit in Denmark or Portugal, due to T1D.
* Age 18 years or above.

Exclusion criteria:

- Severe psychiatric disorder or other conditions deemed to impair the patient's informed consent and participation in the study.

In each country, all subjects from study population 1 will undergo the following assessments at diagnosis of T1D:

1. SARS-Cov-2 antibody measurement.
2. GAD-antibodies (and if necessary islet cell antibodies (IA-2)).
3. HbA1c, fasting blood glucose and fasting C-peptide.
4. Mixed-meal tolerance test (MMTT).
5. Follow-up one year after the diagnosis with HbA1c, fasting blood glucose, fasting C-peptide and MMTT.

Study 2: Epidemiological study 1: In each country, the incidence of SARS-Covid-2 antibodies in study group 1 is compared to the matched control group (Study population 2).

Study 3: Epidemiological study 2: Independently of the above mentioned study, the incidence of newly diagnosed T1D patients in each participant country will be determined by registry data from January 1st 2020 on a monthly basis and compared with newly diagnosed T1D patients from the two previous years (2018 and 2019).

Outcomes

The study will have the following outcomes

Study 1 (clinical study):

Primary outcome: C-peptide AUC of the MMTT at baseline and one year follow-up, for adult T1D patients having SARS-Cov-2 positive vs. negative antibody status.

Secondary outcomes: Fasting glucose, C-peptide, Hba1c at baseline and one year follow-up, for adult T1D patients having SARS-Cov-2 positive vs. negative antibody status.

Study 2 (epidemiological study 1):

Outcome: Proportion of T1D patients having SARS-Cov-2 antibodies, compared to matched controls from the background population, potentially from the national blood banks (1:5 match on age, gender and if possible country region).

Study 3 (epidemiological study 2):

Outcome: Annual and monthly T1D incidence (cases/100.000) during 2020-2022, compared to 2018 and 2019 in Denmark and Portugal.

ELIGIBILITY:
Inclusion Criteria:

* T1D patients diagnosed according to standard practice (including Hba1c, C-peptide, presence of GAD (or islet-cell) antibodies).
* Patient is attending a hospital unit in Denmark or Portugal, due to T1D.
* Age 18 years or above.

Exclusion Criteria:

* Severe psychiatric disorder or other conditions deemed to impair the patient's informed consent and participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All newly diagnosed people with type 1 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Stimulated insulin secretion | One years
  C-peptide AUC of the MMTT at baseline and one year follow-up

SECONDARY OUTCOMES:
HbA1c | One years
  HbA1c measure at one year
Fasting blood glucose | One years
  Fasting blood glucose

CONTACTS AND LOCATIONS:
Overall Officials: Claus B Juhl, Principal Investigator — Esbjerg Hospital - University Hospital of Southern Denmark
Locations (1):
- Hospital of South West Jutland, Esbjerg, Denmark

REFERENCES:
- [Result] Filippi CM, von Herrath MG. Viral trigger for type 1 diabetes: pros and cons. Diabetes. 2008 Nov;57(11):2863-71. doi: 10.2337/db07-1023. No abstract available. PMID 18971433
- [Result] Coleman TJ, Gamble DR, Taylor KW. Diabetes in mice after Coxsackie B 4 virus infection. Br Med J. 1973 Jul 7;3(5870):25-7. doi: 10.1136/bmj.3.5870.25. PMID 4577716
- [Result] Christoffersson G, Flodstrom-Tullberg M. Mouse Models of Virus-Induced Type 1 Diabetes. Methods Mol Biol. 2020;2128:93-105. doi: 10.1007/978-1-0716-0385-7_7. PMID 32180188
- [Result] Stone VM, Hankaniemi MM, Svedin E, Sioofy-Khojine A, Oikarinen S, Hyoty H, Laitinen OH, Hytonen VP, Flodstrom-Tullberg M. A Coxsackievirus B vaccine protects against virus-induced diabetes in an experimental mouse model of type 1 diabetes. Diabetologia. 2018 Feb;61(2):476-481. doi: 10.1007/s00125-017-4492-z. Epub 2017 Nov 18. PMID 29151123
- [Result] Hyoty H, Leon F, Knip M. Developing a vaccine for type 1 diabetes by targeting coxsackievirus B. Expert Rev Vaccines. 2018 Dec;17(12):1071-1083. doi: 10.1080/14760584.2018.1548281. Epub 2018 Nov 29. PMID 30449209
- [Result] Moltchanova EV, Schreier N, Lammi N, Karvonen M. Seasonal variation of diagnosis of Type 1 diabetes mellitus in children worldwide. Diabet Med. 2009 Jul;26(7):673-8. doi: 10.1111/j.1464-5491.2009.02743.x. PMID 19573115
- [Result] Karaoglan M, Eksi F. The Coincidence of Newly Diagnosed Type 1 Diabetes Mellitus with IgM Antibody Positivity to Enteroviruses and Respiratory Tract Viruses. J Diabetes Res. 2018 Aug 16;2018:8475341. doi: 10.1155/2018/8475341. eCollection 2018. PMID 30186878
- [Result] Patterson CC, Gyurus E, Rosenbauer J, Cinek O, Neu A, Schober E, Parslow RC, Joner G, Svensson J, Castell C, Bingley PJ, Schoenle E, Jarosz-Chobot P, Urbonaite B, Rothe U, Krzisnik C, Ionescu-Tirgoviste C, Weets I, Kocova M, Stipancic G, Samardzic M, de Beaufort CE, Green A, Soltesz G, Dahlquist GG. Seasonal variation in month of diagnosis in children with type 1 diabetes registered in 23 European centers during 1989-2008: little short-term influence of sunshine hours or average temperature. Pediatr Diabetes. 2015 Dec;16(8):573-80. doi: 10.1111/pedi.12227. Epub 2014 Oct 15. PMID 25316271
- [Result] Bindom SM, Lazartigues E. The sweeter side of ACE2: physiological evidence for a role in diabetes. Mol Cell Endocrinol. 2009 Apr 29;302(2):193-202. doi: 10.1016/j.mce.2008.09.020. Epub 2008 Oct 1. PMID 18948167
- [Result] Yang JK, Lin SS, Ji XJ, Guo LM. Binding of SARS coronavirus to its receptor damages islets and causes acute diabetes. Acta Diabetol. 2010 Sep;47(3):193-9. doi: 10.1007/s00592-009-0109-4. Epub 2009 Mar 31. PMID 19333547